CLINICAL TRIAL: NCT05768204
Title: Research on the Treatment of Severe Community-acquired Pneumonia in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baoping XU (Other)
Responsible Party: Sponsor-Investigator, Baoping XU, Professor, Beijing Children's Hospital
Organization: Beijing Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCH lung 020
Record Dates: First submitted 2022-12-20; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Severe Pneumonia
Keywords: Severe pneumonia; children; glucocorticoid; Randomized Controlled Trial
MeSH Terms: conditions — Pneumonia | interventions — prednisolone acetate; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Prednisolone, oral, 2 mg/kg.d (maximum dose 60 mg/day), two or three times a day , 5 days.
  Interventions: Drug: Prednisolone Acetate
- Placebo group (Placebo Comparator): The same amount of placebo was taken orally as the trial for 5 days
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Prednisolone Acetate — The experimental group took prednisolone acetate which is a kind of oral glucocorticoid.
  Other Names: Prednisolone
  Arms: Experimental group
Other: placebo — A placebo consistent in appearance with the prednisolone acetate.
  Arms: Placebo group

SUMMARY:
The need for glucocorticoid therapy in children with severe community-acquired pneumonia in the acute phase of the disease remains unclear. The implementation of this study could provide strong evidence on the need for adjuvant glucose therapy in children with severe community-acquired pneumonia.

DETAILED DESCRIPTION:
The use of glucocorticoid for severe community-acquired pneumonia in children is still controversial in clinic. There is still a lack of high quality clinical research results in this field. That's the purpose of this study. The study used oral glucocorticoids and placebos. It was a multicenter clinical study involving 160 people. The enrolled subjects were treated for 5 days after basic assessment, and the use of experimental drugs and changes in clinical manifestations and laboratory examination were strictly recorded. The possible adverse hormonal reactions such as hyperglycemia, hypertension and gastrointestinal ulcer bleeding should be closely monitored and appropriate treatment measures should be taken in time. Subject will be allowed to terminate the test if necessary. Record and discuss similar events. The double blind principle is strictly observed during the experiment to ensure the authenticity and reliability of the experimental data.

ELIGIBILITY:
Inclusion Criteria:

1. 1 month-< 18 years old.
2. Clinical diagnosis of community-acquired pneumonia (fever, cough, sputum, chest pain, dyspnea, abnormal breath sounds in the lungs, imaging pneumonia changes).
3. Meet any of the following:

   * (1) the general condition is very poor;
   * (2) refusal to eat or dehydration;
   * (3) Significantly increased respiratory rate (70 times/min > infants, 50 times/min for older children>);
   * (4) dyspnea (three concave sign, moaning, nasal flapping)
   * (5) hypoxemia (cyanosis, transcutaneous oxygen saturation< 92% (not oxygenated));
   * (6) Pulmonary infiltration≥ 2/3 lung or multilobar infiltration;
   * (7) There is a pleural effusion;
   * (8) Extrapulmonary complications

Exclusion Criteria:

1. Systemic corticosteroids have been used to treat pneumonia before admission.
2. Use systemic glucocorticoids within 3 months before admission.
3. Hospital-acquired pneumonia.
4. Children with history of tuberculosis, branch expansion, tumors, immune deficiency, congenital heart, chronic pulmonary heart disease, kidney disease, severe malnutrition, recurrent respiratory infections, congenital bronchopulmonary dysplasia (BPD) and other underlying diseases.
5. Unconscious, need endotracheal intubation, children admitted to ICU.
6. Those who are allergic to the drugs or their preparation components involved in the study.
7. Those with hormonal contraindications: hypertension, diabetes, active peptic ulcer, adrenal hyperfunction, corneal ulcer, increased intraocular pressure, severe psychosis.
8. There is a current infection that is difficult to control with antibacterial drugs.
9. Children who are participating in other clinical trials.
10. The investigator believes that it is not suitable to participate in the study.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
the rate of early treatment success | third day
  temperature is normal, clinical manifestations are significantly improved, pulmonary signs are significantly improved or disappeared, and white blood cell\C reactive protein\procalcitonin returns to normal

CONTACTS AND LOCATIONS:
Overall Officials: Baoping Xu, Study Director — Beijing Children's Hospital
Locations (3):
- China (3):
  - Baoding Children's Hospital, Baoding
  - Beijing Children's Hospital, Beijing
  - Beijing Fangshan District Health Care Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No